CLINICAL TRIAL: NCT02039882
Title: Point of Care (POC) Biomarkers of Ischemia
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM15114
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Acute Coronary Syndrome (ACS); Percutaneous Coronary Intervention PCI; Normals; Myocardial Infarction MI; Point of Care POC; Hypoxanthine; Inosine; HPLC High Pressure Liquid Chromatography
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood, Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controls/Normals: control subjects without known cardiac disease, age ± 5 years and sex matched
- Acute Coronary Syndrome requiring Percutaneous Intervention: Subjects presenting to ER with Acute chest pain requiring cardiac catheterization
- Acute Coronary Syndrome, no intervention: Acute Coronary Syndrome, not requiring Percutaneous intervention

SUMMARY:
Acute coronary syndrome is defined as myocardial infarction or ischemia as evidenced by significant coronary artery disease on cardiac catheterization/revascularization or reversible defect seen on stress test. Each year approximately 8-10 million patients undergo an emergency department evaluation for possible acute coronary syndrome (ACS) in the United States Up to 8%of patients who have myocardial infarction (MI) are inadvertently discharged. Unnecessary admissions for presumed myocardial disease result in health care costs that are estimated to exceed 5 billion dollars annually Currently, the cardiac biomarkers troponin and Creatine phosphokinase (CPK-MB), in conjunction with ECG changes are used to evaluate a patient routinely for ACS. However, these tests have limitations for identifying most patients who have ACS in a rapid fashion. Purine molecules such as inosine and hypoxanthine and have been shown to also be biomarkers of acute MI. High pressure liquid chromatography (HPLC) is the traditional method of analysis of these purines. The HPLC method however requires hours to assess biomarkers, as do the more traditionally used troponin and CK-MB methods.

Recently, the investigator has developed a rapid chemo luminescence method for detecting purine biomarkers. This modality can provide an expeditious (requires less than 4 minutes to complete analysis), bedside method of analysis for ACS through routinely acquired blood samples. In this study the investigator will compare the results of the chemo luminescence method with the gold standard HPLC method, and results of the traditional cardiac markers troponin and Creatine phosphokinase (CK-MB) in patients undergoing an evaluation for ACS. Details of noninvasive and invasive cardiac assessments performed as part of the routine evaluation by the clinician for myocardial assessment and intervention in conjunction with biomarker assessment will be obtained. The investigator hypothesize that the rapid chemo luminescence biomarker assessment will identify patients with ACS faster than traditional diagnostic methods.

The goal of this study is to assess the role of rapid assessment of purine biomarkers in identifying patients who may have ACS.

DETAILED DESCRIPTION:
Fifty patients presenting for evaluation of ACS (acute coronary syndrome) in the hospital emergency department (ED) will be studied and 50 control subjects without known cardiac disease that are age ± 5years and sex matched. Pregnant women, children and prisoners as well as individuals with hemoglobin less than 9 g/dL will be excluded. Blood will be drawn to analyze for the biomarkers inosine, and hypoxanthine at the time standard of care biomarker troponin is sampled. The levels of the biomarkers inosine and hypoxanthine will be measured by our research laboratory, using LC/mass spectrometry(MS) and luminescence methodologies. Troponin levels will be measured as standard of care in the routine fashion by the hospital laboratory (CLIA accredited) at Virginia Commonwealth University Medical Center. Demographic and clinical information will be obtained and the clinical course followed. EKG data, cardiac angiography and other cardiac assessment data (e.g. ECHO, rest and stress myocardial perfusion imaging) that is performed as part of the standard of care evaluation will be collected and evaluated. A maximum of (6) 10 ml blood samples (heparin anticoagulant) for analysis will be drawn throughout the hospitalization.

Twenty Five patients presenting with ACS not requiring an immediate (PCI) Percutaneous Coronary Intervention: will have samples drawn at 0, 3 and 6 hours after vascular access has been acquired. Blood samples for analysis as standard of care for troponin are at 0, 3 and 6 hours.

Twenty Five patients presenting with ACS requiring an immediate PCI Percutaneous Coronary Intervention will have blood samples drawn at time 0, immediately after intervention, 1, 3 and 6 hours. Troponin samples will be acquired and analyzed as per routine practice (time 0, 3, 6 hour) and (2) additional troponin samples will be collected (after reperfusion and 1 hour). The analytical costs of these (2) samples will be charged to the department of Nephrology.

Fifty age ± 5years and sex matched control subjects without known cardiac disease will have timed blood samples drawn at 0, 3 and 6 hours. These samples will be analyzed for troponin, inosine and hypoxanthine.

These patient samples will serve as the control group. Control subjects will be recruited from the Virginia Commonwealth University Health Systems.

Due to the acute nature of the patients presenting with chest pain, a 10 ml sample of blood will be drawn at the time of the first routine blood draw for clinical purposes and the samples reserved until patient consent can be discussed. If patient consents to participate the sample will be retained and added to other study samples. If declined the sample will be discarded.

Hypoxanthine and Inosine levels will be measured by LC/MS (mass spectrometry) methods. Luminescence technology used will be utilizing Lumistar Optima Microplate Reader. Analysis of samples will be completed in batches throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting for evaluation of ACS (acute coronary syndrome) in the hospital emergency department (ED) control subjects without known cardiac disease that are age ± 5 years and sex matched to subjects with Acute coronary Syndrome

* Men and Women over age of 18
* Women who are not pregnant
* Subject who are not prisoners
* Hemoglobin greater than or equal to 9mg/dl
* Subjects who speak english
* Subjects 18 years of age or older

Exclusion Criteria:

Men and Women under the age of 18 Women who are pregnant Subject who are prisoners Subjects who do not speak English Individuals with hemoglobin less than 9 g/dL Control subjects with known heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty total patients presenting for evaluation of ACS (acute coronary syndrome) in the hospital emergency department (ED) at Virginia Commonwealth University Health Systems, Twenty five Patents requiring percutaneous Intervention, Twenty five patients not requiring intervention Fifty control subject from Virginia Commonwealth University Health Systems without known cardiac disease that are age ± 5years and sex matched from
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12-15 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
Point of care Biomarkers of Ischemia Correlation | one year
  correlation of biomarkers of inosine and hypoxanthine measurements using rapid chemoluminescence method with HPLC quantitation. Subjects with ACS not requiring an immediate (PCI) Percutaneous Coronary Intervention: will have samples drawn at 0, 3 and 6 hours after vascular access has been acquired. Blood samples for analysis as standard of care for troponin are at 0, 3 and 6 hours. ACS requiring an immediate PCI Percutaneous Coronary Intervention will have blood samples drawn at time 0, immediately after intervention, 1, 3 and 6 hours. Troponin samples will be acquired and analyzed as per routine practice (time 0, 3, 6 hour) and (2) additional troponin samples will be collected (after reperfusion and 1 hour).

SECONDARY OUTCOMES:
Point of Care Biomarkers of Ischemia Comparison | one year
  Investigator will compare measurements of inosine and hypoxanthine with traditional markers of MI, Subjects with ACS not requiring an immediate (PCI) Percutaneous Coronary Intervention: will have samples drawn at 0, 3 and 6 hours after vascular access has been acquired. Blood samples for analysis as standard of care for troponin are at 0, 3 and 6 hours. ACS requiring an immediate PCI Percutaneous Coronary Intervention will have blood samples drawn at time 0, immediately after intervention, 1, 3 and 6 hours. Troponin samples will be acquired and analyzed as per routine practice (time 0, 3, 6 hour) and (2) additional troponin samples will be collected (after reperfusion and 1 hour).

CONTACTS AND LOCATIONS:
Overall Officials: Todd Gehr, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealtlh University Health Systems, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided